CLINICAL TRIAL: NCT03498963
Title: Early Detection by Molecular Biology Technique of Pathogens Responsible for Respiratory Infections Associated With Drownings in Seawater: Pilot Study at the CHU de Nice
Brief Title: Pathogens Responsible for Respiratory Infections Associated With Drowning in Seawater
Acronym: APIR-NOY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-AOIP-03
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Drowning
MeSH Terms: conditions — Drowning | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bronchoalveolar lavage (Other)
  Interventions: Procedure: bronchoalveolar lavage

INTERVENTIONS:
Procedure: bronchoalveolar lavage — Carrying out a bronchoalveolar lavage (BAL) within 24 hours after admission to intensive care with analysis on standard and specific culture media of environmental germs, carrying out antibiograms, DNA extraction, amplification by universal 16 and 18S rDNA primers followed by high flow sequencing and phylogenetic analysis of pathogens found. Comparison of these results with the same analyses performed on seawater samples taken near the drowning site and during a new AML at 72h for patients still intubated and showing signs of pneumonia in order to determine if the pathogens detected at the entrance persist and are present in the environment.

SUMMARY:
Little data is currently available on the type of pathogen responsible for respiratory infections following drowning. Many environmental germs present in seawater are described as difficult to culture on standard media but are potentially pathogenic. Even using specific culture media nearly 90% of the bacteria present in the water remain non-cultivable. The use of 16S and 18S rDNA amplification followed by high throughput sequencing on respiratory samples could allow us to objectify these bacteria potentially involved in the physiopathological process secondary to drowning and thus improve their overall management.

Carrying out a bronchoalveolar lavage (BAL) within 24 hours after admission to intensive care with analysis on standard and specific culture media of environmental germs, carrying out antibiograms, DNA extraction, amplification by universal 16 and 18S rDNA primers followed by high flow sequencing and phylogenetic analysis of pathogens found. Comparison of these results with the same analyses performed on seawater samples taken near the drowning site and during a new AML at 72h for patients still intubated and showing signs of pneumonia in order to determine if the pathogens detected at the entrance persist and are present in the environment.

AML at the patient's entrance, on day 3 and environmental sampling in the drowning environment within 24 hours. Standard and specific bacteriological analyses with molecular biology techniques (amplification 16 and 18S rDNA) carried out at Pr RUIMY's laboratory (Nice University Hospital) sequencing on INRA's Toulouse genomics platform. Phylogenetic data capture and analysis at IRCAN (Bioinformatics, Croce Olivier). Patient follow-up until resuscitation discharge.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* hospitalized in intensive care for severe drowning in sea water (Spilzman stage 5 or 6) (4)
* intubated within 24 hours of admission or before admission to intensive care
* affiliated to social security

Exclusion Criteria:

* patients under guardianship, trusteeship or detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
presence of potentially pathogenic seawater germs not detected by standard cultures and found in the drowning environment. | 3 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Frejus hospital, Fréjus
  - university hospital of Nice, Nice

IPD SHARING:
Plan to Share IPD: No